CLINICAL TRIAL: NCT02215200
Title: Antithymocyte Globulin (ATG) and Pegylated Granulocyte Colony Stimulating Factor (GCSF) in New Onset Type 1 Diabetes
Brief Title: ATG-GCSF in New Onset Type 1 Diabetes
Acronym: ATG-GCSF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Research Resources (NCRR) (NIH); Juvenile Diabetes Research Foundation (Other); American Diabetes Association (Other); Sanofi (Industry); The Leona M. and Harry B. Helmsley Charitable Trust (Other); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATG-GCSF (IND); Type 1 Diabetes TrialNet (Other: Type 1 Diabetes TrialNet); TN19 (Other: Type 1 Diabetes TrialNet); UC4DK106993 (NIH); UC4DK117009 (NIH)
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes TrialNet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; thymoglobulin; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Anti-Thymocyte Globulin (ATG) and Placebo (Experimental): Anti-Thymocyte Globulin (ATG)/Placebo: Anti-Thymocyte Globulin (ATG) will be administered at a dose of 2.5mg/kg as two divided IV infusions of 0.5mg/kg and 2mg/kg. First dose (0.5mg/kg) will be infused over a minimum of 12 hours, and the second dose (2mg/kg) over a minimum of 8 hours. The second dose should be given no less than 12 and no more than 24 hours after the previous dose.
  Placebo(for GCSF) treatment will begin 6 hours after completion of the ATG. Placebo will be given subcutaneously every 2 weeks for a total of 6 doses
  Interventions: Drug: Anti-Thymocyte Globulin (ATG); Drug: Placebo (for GCSF)
- ATG plus Granulocyte colony stimulating factor (GCSF) (Experimental): Granulocyte colony stimulating factor (GCSF) is supplied in 0.6 mL prefilled syringes for subcutaneous injection. Each syringe contains 6 mg GCSF (based on protein weight), in a sterile, clear, colorless, preservative-free solution (pH 4.0) containing acetate (0.35 mg), sorbitol (30.0 mg), polysorbate 20 (0.02 mg), and sodium (0.02 mg) in water for injection, U.S. Pharmacopeial Convention (USP). The standard 6mg dose will be given with the exception of subjects who weigh less than 45 kg.
  GCSF treatment will begin 6 hours after completion of the ATG / Placebo. GCSF will be given subcutaneously every 2 weeks for a total of 6 doses
  Interventions: Drug: Anti-Thymocyte Globulin (ATG); Drug: Granulocyte colony stimulating factor (GCSF)
- Placebo (Placebo Comparator): Placebo for ATG will be administered by IV infusion in 2 doses. Placebo for GCSF will be administered subcutaneously every 2 weeks for a total of 6 doses
  Interventions: Drug: Placebo (for ATG); Drug: Placebo (for GCSF)

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin (ATG) — Thymoglobulin
  Other Names: Thymoglobulin
  Arms: ATG plus Granulocyte colony stimulating factor (GCSF); Anti-Thymocyte Globulin (ATG) and Placebo
Drug: Granulocyte colony stimulating factor (GCSF) — Granulocyte colony stimulating factor (GCSF)
  Other Names: Neulasta
  Arms: ATG plus Granulocyte colony stimulating factor (GCSF)
Drug: Placebo (for ATG) — Normal saline administered by IV infusion to mimic ATG
  Arms: Placebo
Drug: Placebo (for GCSF) — Placebo prepared to mimic 6mg subcutaneous injection of GCSF
  Arms: Anti-Thymocyte Globulin (ATG) and Placebo; Placebo

SUMMARY:
This is a three-arm, 1:1:1 randomized, placebo controlled, double- blinded trial in which at least 28 subjects will receive active Anti-Thymocyte Globulin and Granulocyte colony-stimulating factor (ATG-GCSF), at least 28 subjects will receive ATG alone and at least 28 subjects will receive placebo alone within 100 days from diagnosis of Type 1 Diabetes (T1D).

The primary objective of the study will be to determine the safety and ability of low dose ATG plus GCSF and low dose ATG alone to retain/enhance C-peptide production in new onset T1D patients demonstrating residual beta cell function.

DETAILED DESCRIPTION:
The primary statistical hypothesis to be assessed in the study is whether the 2 hour area under the curve (change in baseline to 12 months) in residual beta cell function (C-peptide) will differ between those treated with ATG and GCSF or ATG alone as compared with placebo.

The study will also examine the effect of the proposed treatments on surrogate markers for immunologic and metabolic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must be > 12 years < 46
* Must have a diagnosis of T1D for less than 100 days at randomization
* Willing to provide Informed Consent or have a parent or legal guardian provide informed consent if the subject is <18 years of age
* Positive for at least one islet cell autoantibody; glutamic acid decarboxylase 65 (GAD65A), Insulin micro IAA (mIAA), if obtained within 10 days of the onset of insulin therapy, islet antigen 2 (IA-2A), Islet Cell Antigen (ICA), or zinc transporter 8 (ZnT8A)
* Must have stimulated C-peptide levels = 0.2 pmol/ml measured during a mixed meal tolerance test (MMTT) conducted at least 21 days from diagnosis of diabetes and within one month (37 days) of randomization
* Must be Epstein-Barr virus (EBV PCR) negative within two weeks of randomization if EBV seronegative at screening
* Be at least 6 weeks from last live immunization
* Participants are required to receive killed influenza vaccination at least 2 weeks prior to randomization when vaccine for the current or upcoming flu season is available
* Be willing to forgo vaccines during the treatment period and for 3 months following last dose of study drug
* Be willing to comply with intensive diabetes management

Exclusion Criteria:

* Be immunodeficient or have clinically significant chronic lymphopenia: (Leukopenia (< 3,000 leukocytes /µL), neutropenia (<1,500 neutrophils/µL), lymphopenia (<800 lymphocytes/µL), or thrombocytopenia (<100,000 platelets/µL).
* Have active signs or symptoms of acute infection at the time of randomization
* Have evidence of prior or current tuberculosis infection as assessed by purified protein derivative (PPD), interferon gamma release assay (IGRA) or by history
* Be currently pregnant or lactating, or anticipate getting pregnant within the two year study period
* Require use of other immunosuppressive agents including chronic use of systemic steroids
* Have evidence of current or past human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection
* Have any complicating medical issues or abnormal clinical laboratory results that may interfere with study conduct, or cause increased risk to include pre-existing cardiac disease, chronic obstructive pulmonary disease (COPD), sickle cell disease, neurological, or blood count abnormalities
* Have a history of malignancies other than skin
* Evidence of liver dysfunction with aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 3 times the upper limits of normal
* Evidence of renal dysfunction with creatinine greater than 1.5 times the upper limit of normal
* Vaccination with a live virus within the last 6 weeks
* Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within prior 7 days of screening
* Active participation in another T1D treatment study in the previous 30 days
* Prior treatment with abatacept or anti-cd3
* Known allergy to GCSF or ATG
* Prior treatment with ATG or known allergy to rabbit derived products
* Any condition that in the investigator's opinion may adversely affect study participation or may compromise the study results

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 89 (Actual)
Dates: Start 2014-12; Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Haller, M.D., Principal Investigator — University of Florida
Locations (13):
- United States (13):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida Diabetes Center, Tampa, Florida
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University-Naomi Berrie Diabetes Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Eskind Diabetes Clinic, Nashville, Tennessee
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository
Supporting Information: Study Protocol, CSR, Analytic Code
URL: https://repository.niddk.nih.gov/studies/TN19_ATG_GCSF/?query=tn19

REFERENCES:
- [Derived] Jacobsen LM, Diggins K, Blanchfield L, McNichols J, Perry DJ, Brant J, Dong X, Bacher R, Gersuk VH, Schatz DA, Atkinson MA, Mathews CE, Haller MJ, Long SA, Linsley PS, Brusko TM. Responders to low-dose ATG induce CD4+ T cell exhaustion in type 1 diabetes. JCI Insight. 2023 Aug 22;8(16):e161812. doi: 10.1172/jci.insight.161812. PMID 37432736
- [Derived] Haller MJ, Long SA, Blanchfield JL, Schatz DA, Skyler JS, Krischer JP, Bundy BN, Geyer SM, Warnock MV, Miller JL, Atkinson MA, Becker DJ, Baidal DA, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Herold KC, Marks JB, Moran A, Rodriguez H, Russell WE, Wilson DM, Greenbaum CJ; Type 1 Diabetes TrialNet ATG-GCSF Study Group. Low-Dose Anti-Thymocyte Globulin Preserves C-Peptide, Reduces HbA1c, and Increases Regulatory to Conventional T-Cell Ratios in New-Onset Type 1 Diabetes: Two-Year Clinical Trial Data. Diabetes. 2019 Jun;68(6):1267-1276. doi: 10.2337/db19-0057. Epub 2019 Apr 9. PMID 30967424
- [Derived] Haller MJ, Schatz DA, Skyler JS, Krischer JP, Bundy BN, Miller JL, Atkinson MA, Becker DJ, Baidal D, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Herold KC, Marks JB, Moran A, Rodriguez H, Russell W, Wilson DM, Greenbaum CJ; Type 1 Diabetes TrialNet ATG-GCSF Study Group. Low-Dose Anti-Thymocyte Globulin (ATG) Preserves beta-Cell Function and Improves HbA1c in New-Onset Type 1 Diabetes. Diabetes Care. 2018 Sep;41(9):1917-1925. doi: 10.2337/dc18-0494. Epub 2018 Jul 16. PMID 30012675
- See also: Type 1 Diabetes TrialNet — http://www.diabetestrialnet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Anti-Thymocyte Globulin (ATG) and Placebo: Anti-Thymocyte Globulin (ATG)/Placebo: Anti-Thymocyte Globulin (ATG) will be administered at a dose of 2.5mg/kg as two divided IV infusions of 0.5mg/kg and 2mg/kg. First dose (0.5mg/kg) will be infused over a minimum of 12 hours, and the second dose (2mg/kg) over a minimum of 8 hours. The second dose should be given no less than 12 and no more than 24 hours after the previous dose.
  Placebo(for GCSF) treatment will begin 6 hours after completion of the ATG. Placebo will be given subcutaneously every 2 weeks for a total of 6 doses
  Anti-Thymocyte Globulin (ATG): Thymoglobulin
  Placebo (for GCSF): Placebo prepared to mimic 6mg subcutaneous injection of GCSF
- ATG Plus Granulocyte Colony Stimulating Factor (GCSF): Granulocyte colony stimulating factor (GCSF) is supplied in 0.6 mL prefilled syringes for subcutaneous injection. Each syringe contains 6 mg GCSF (based on protein weight), in a sterile, clear, colorless, preservative-free solution (pH 4.0) containing acetate (0.35 mg), sorbitol (30.0 mg), polysorbate 20 (0.02 mg), and sodium (0.02 mg) in water for injection, U.S. Pharmacopeial Convention (USP). The standard 6mg dose will be given with the exception of subjects who weigh less than 45 kg.
  GCSF treatment will begin 6 hours after completion of the ATG / Placebo. GCSF will be given subcutaneously every 2 weeks for a total of 6 doses
  Anti-Thymocyte Globulin (ATG): Thymoglobulin
  Granulocyte colony stimulating factor (GCSF): Granulocyte colony stimulating factor (GCSF)
Period: Overall Study
Arm/Group | Anti-Thymocyte Globulin (ATG) and Placebo | ATG Plus Granulocyte Colony Stimulating Factor (GCSF) | Placebo
Started | 29 | 29 | 31
Completed | 29 | 28 | 30
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-Thymocyte Globulin (ATG) and Placebo | ATG Plus Granulocyte Colony Stimulating Factor (GCSF) | Placebo | Total
Number analyzed (Participants) | 29 | 29 | 31 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17.2 (5) | 18.1 (6.9) | 16.9 (4.6) | 17.4 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 14 | 39
  Male | 16 | 17 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 28 | 27 | 30 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 28 | 29 | 29 | 86
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 31 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Under the Stimulated C-peptide Curve From Baseline to 12 Months.
Description: The C-peptide 2 hour area under the curve (AUC) mean is calculated at baseline and 12 months and measured in nmol/L. The calculation for the concentration of c-peptide is a weighted average of the 6 timed measurements of c-peptide in nano-moles/Liter. We try to distinguish this calculation from the AUC by referring to it as the "AUC mean" and may be expressed algebraically as the AUC/(120 min.); thus, the units are the same as the y-axis").
Time Frame: -10, 0 15, 30, 60, 90, and 120 minutes post-dose at baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Anti-Thymocyte Globulin (ATG) and Placebo | ATG Plus Granulocyte Colony Stimulating Factor (GCSF) | Placebo
Number analyzed (Participants) | 29 | 28 | 30
nmol/L | 0.528 [0.435 to 0.627] | 0.646 [0.547 to 0.750] | 0.406 [0.324 to 0.494]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year.
Description: Adverse events were defined using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Anti-Thymocyte Globulin (ATG) and Placebo | ATG Plus Granulocyte Colony Stimulating Factor (GCSF) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 28/29 | 29/29 | 8/31
Other Adverse Events (participants affected / at risk) | 28/29 | 29/29 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-Thymocyte Globulin (ATG) and Placebo (N=29) | ATG Plus Granulocyte Colony Stimulating Factor (GCSF) (N=29) | Placebo (N=31)
All immune system disorders (Immune system disorders) | 12 (14) | 15 (15) | 0 (0)
CD4 lymphocyte decrease or other (Blood and lymphatic system disorders) | 18 (24) | 17 (23) | 0 (0)
General Disorders and administration (General disorders) | 2 (4) | 1 (1) | 1 (1)
Endocrine Disorders (Endocrine disorders) | 0 (0) | 0 (0) | 1 (5)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Psychiatric Disorders (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2)
Neoplasms: benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-Thymocyte Globulin (ATG) and Placebo (N=29) | ATG Plus Granulocyte Colony Stimulating Factor (GCSF) (N=29) | Placebo (N=31)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 5 (6) | 7 (10) | 4 (7)
All Immune system disorders (Immune system disorders) | 21 (33) | 23 (38) | 0 (0)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 10 (14) | 3 (3) | 5 (6)
CD4 lymphocyte decrease or other (Blood and lymphatic system disorders) | 21 (42) | 22 (43) | 3 (4)
General Disorders and administration (General disorders) | 7 (16) | 8 (18) | 1 (1)
Endocrine Disorders (Endocrine disorders) | 1 (1) | 1 (1) | 3 (7)
Infections and infestations (Infections and infestations) | 9 (14) | 7 (9) | 9 (16)
Gastrointestinal Disorders (Gastrointestinal disorders) | 5 (7) | 3 (5) | 6 (6)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Psychiatric Disorders (Psychiatric disorders) | 2 (7) | 1 (1) | 0 (0)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 1 (4) | 2 (2) | 5 (5)
Nervous system disorders (Nervous system disorders) | 4 (4) | 4 (11) | 2 (5)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (7) | 2 (4) | 4 (4)
Vascular Disorders (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Neoplasms: benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Respiratory, thoracic, and mediastinal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 1 (1)
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02215200/Prot_000.pdf
  • Informed Consent Form (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02215200/ICF_001.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT02215200/SAP_002.pdf